CLINICAL TRIAL: NCT02175056
Title: A Dose-Block Randomized, Placebo Controlled (Double-blind), Active Controlled(Open-label), Dose-escalation Study to Investigate the Tolerability, and Pharmacokinetics/Pharmacodynamics of HL2351 After a Single Subcutaneous Administration in Healthy Male Subjects
Brief Title: A Dose-Block Randomized, Placebo Controlled (Double-blind), Active Controlled(Open-label), Dose-escalation Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HL_C101
Record Dates: First submitted 2014-06-17; First posted 2014-06-26 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Healthy Volunteers
Keywords: First In Human; CAPS, SoJIA, AOSD, Bechet Disease, Rheumatoid arthritis
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes; Arthritis, Rheumatoid | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- HL2351 (Experimental): 1, 2, 4, 8, 12 mg/kg (SC) / Single-Dose
  Interventions: Biological: HL2351
- Placebo (Placebo Comparator): 1, 2, 4, 8, 12 mg/kg (SC) / Single-Dose
  Interventions: Biological: HL2351
- Kineret(Anakinra) (Active Comparator): 100 mg (SC) / Single-Dose
  Interventions: Biological: Kineret(Anakinra)

INTERVENTIONS:
Biological: HL2351 — Dose-escalation For 5 level dose groups A ~ E(each 1, 2, 4, 8, 12mg/kg), 10 subjects (8 for the study drug and 2 for placebo) are randomized to each dose group, and the study drug or placebo is subcutaneously administered for the relevant dose group.
  Arms: HL2351; Placebo
Biological: Kineret(Anakinra) — Active comparator(group F) is implemented in parallel with dose groups A~E in an open-label manner and 8 subjects subcutaneously administer Kineret® 100 mg.
  Arms: Kineret(Anakinra)

SUMMARY:
The study design of this trial is a Dose-Block Randomized, Placebo controlled (Double-blind), Active Controlled(Open-label), Dose-escalation.

DETAILED DESCRIPTION:
* Extended in vivo half-life of HL2351 is also anticipated to provide improved therapeutic efficacy based on sustained maintenance of an effective concentration.
* A safety concern may be addressed by utilizing IL-1Ra that is being used after getting approval by the EMA and the US FDA and known to be relatively safe, and the Fc fusion technology that has been already applied to various therapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy adult man aged between 20 and 45 years (inclusive) at screening
2. Weight between 55 and 90 kg (inclusive) and the body mass index(BMI) between 18.0 and 27.0 (inclusive)

   * BMI(kg/m2) = Body weight (kg)/{height (m)}2
3. Voluntary consent to participation in this study and signature on the IRB-approved informed consent form after being explained about characteristics of this clinical study, prior to any screening test

Exclusion Criteria:

1. Current or history of a clinically significant hepatic, renal, neurological, immunological, respiratory or endocrine disease or hematological or oncological disease, cardiovascular disease or psychiatric disease (mood disorder or compulsive disorder, etc.) (in case of a hepatic disease, a hepatitis virus-infected subject may be also included)
2. Hypersensitivity to a drug (aspirin or antibiotics, etc.) or past history of clinically significant hypersensitivity
3. In sitting vital signs measured after resting for 3 min or more, systolic blood pressure of <90mmHg or >150mmHg, or diastolic blood pressure of <60mmHg or >100 mmHg
4. Past history of drug abuse or positive urine drug screening results
5. Use of any prescription medicine or oriental medicine within 2 weeks or use of any over-the-counter(OTC) medication or vitamin preparation within 1 week prior to the scheduled first dose (however, a subject may be included if other conditions are satisfied, at the discretion of the investigator)
6. Participation in another clinical study and administration of a drug within 3 months prior to the scheduled first dose (from the dosing day)
7. Whole blood donation within 2 months or apheresis within 1 month prior to the scheduled first dose, or transfusion within 1 month prior to the first dose
8. A habitual drinker (>21 units/week, 1 unit = 10 g of pure alcohol) or a person who cannot abstain from alcohol consumption during hospitalization
9. A smoker of 10 cigarettes/day on average over the past 3 months or a person who cannot abstain from smoking during hospitalization
10. A person who is planning to get pregnant during the study or who cannot practice acceptable contraception (example: surgical sterilization of a subject or a partner, intrauterine device used by a partner, barrier contraception, diaphragm or condom used in combination) even if not planning to get pregnant
11. Notable prolongation of the QT/QTcb interval at screening (e.g., repeated confirmation of QTcb interval > 450 ms)
12. Confirmed history of a risk factor for TdP (e.g., heart failure, hypokalemia, family history of a long QT syndrome)
13. Chronic, uncontrolled or symptomatic inflammatory disease (e.g., rheumatoid arthritis, systemic lupus erythematosis)
14. Pyrexia of ≥38°C within 1 week prior to administration of the investigational product
15. Past history of tuberculosis infection and/or positive Quantiferon TB-Gold test results at screening
16. A person who had participated in this study and received the investigational product
17. A person who is otherwise determined as not eligible for clinical study participation by the investigator due to other reasons including clinical laboratory test results

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Tolerability as measured by the occurrence of Adverse Events | 29 days
  Adverse Events after single subcutaneous dose of HL2351
  : check Day -1, 1, 2, 3, 4, 5, 7, 11, 15, 22, 29
Tolerability as measured by Physical Examination, Vital Signs and Safety Laboratory Tests | 29 days
  Changes from baseline in physical examination, vital signs, ECG, clinical laboratory tests (routine hematology, routine chemistry, blood coagulation and urinalysis) after single subcutaneous dose of HL2351
Tolerability as measured by the occurrence of Local Toxicity | 4 days
  Local Toxicity after single subcutaneous dose of HL2351
  : check Day 1, 2, 4
Tolerability as measured by Cytokine Laboratory Test | 4 days
  Cytokine Laboratory Test after single subcutaneous dose of HL2351
  : check Day 1, 2, 4
Pharmacokinetics of HL2351: Maximum plasma concentration(Cmax) | 29 days
  To assess pharmacokinetics after single subcutaneous injection of HL2351
Pharmacokinetics of HL2351: Area under plasma drug concentration-time curve [AUC(0-last), AUCinf] | 29 days
  To assess pharmacokinetics after single subcutaneous injection of HL2351
Pharmacokinetics of HL2351: Time of maximum concentration(Tmax) | 29 days
  To assess pharmacokinetics after single subcutaneous injection of HL2351
Pharmacokinetics of HL2351: Elimination half-life(T1/2) | 29 days
  To assess pharmacokinetics after single subcutaneous injection of HL2351
Pharmacokinetics of HL2351: Apparent Clearance(CL/F) | 29 days
  To assess pharmacokinetics after single subcutaneous injection of HL2351
Pharmacokinetics of HL2351: Apparent Volume of Distribution(Vz/F) | 29 days
  To assess pharmacokinetics after single subcutaneous injection of HL2351
Pharmacokinetics of HL2351: Mean Residence Time (MRT) | 29 days
  To assess pharmacokinetics after single subcutaneous injection of HL2351
Pharmacodynamics of HL2351: IL-6 inhibition assay | 7 days
  To assess the pharmacodynamic dose-response relationship after single subcutaneous injection of HL2351 IL-6 inhibition assay: AUEClast, Emax

SECONDARY OUTCOMES:
Immunogenicity of HL2351: Anti-drug Antibody | Day 1, Day 29
  To assess immunogenicity after single subcutaneous injection of HL2351
Tolerability in comparison with Kineret(Anakinra): measured by the occurrence of Adverse Events | 3 days
  To explore tolerability in comparison with subcutaneous administration of a positive comparator, Kineret(Anakinra)
Tolerability in comparison with Kineret(Anakinra): measured by Physical Examination, Vital Signs and Safety Laboratory Tests | 3 days
  To explore tolerability in comparison with subcutaneous administration of a positive comparator, Kineret(Anakinra)
Tolerability in comparison with Kineret(Anakinra): measured by the occurrence of Local Toxicity | 3 days
  To explore tolerability in comparison with subcutaneous administration of a positive comparator, Kineret(Anakinra)
Tolerability in comparison with Kineret(Anakinra): measured by Cytokine Laboratory Test | 3 days
  To explore tolerability in comparison with subcutaneous administration of a positive comparator, Kineret(Anakinra)
Pharmacokinetics in comparison with Kineret(Anakinra): Maximum plasma concentration | 3 days
  To explore pharmacokinetics in comparison with subcutaneous administration of a positive comparator, Kineret(Anakinra)
Pharmacokinetics in comparison with Kineret(Anakinra): Area under plasma drug concentration-time curve [AUC(0-last), AUCinf] | 3 days
  To explore pharmacokinetics in comparison with subcutaneous administration of a positive comparator, Kineret(Anakinra)
Pharmacokinetics in comparison with Kineret(Anakinra): Time of maximum concentration(Tmax) | 3 days
  To explore pharmacokinetics in comparison with subcutaneous administration of a positive comparator, Kineret(Anakinra)
Pharmacokinetics in comparison with Kineret(Anakinra): Elimination half-life(T1/2) | 3 days
  To explore pharmacokinetics in comparison with subcutaneous administration of a positive comparator, Kineret(Anakinra)
Pharmacokinetics in comparison with Kineret(Anakinra): Apparent Clearance(CL/F) | 3 days
  To explore pharmacokinetics in comparison with subcutaneous administration of a positive comparator, Kineret(Anakinra)
Pharmacokinetics in comparison with Kineret(Anakinra): Apparent Volume of Distribution(Vz/F) | 3 days
  To explore pharmacokinetics in comparison with subcutaneous administration of a positive comparator, Kineret(Anakinra)
Pharmacokinetics in comparison with Kineret(Anakinra): Mean Residence Time (MRT) | 3 days
  To explore pharmacokinetics in comparison with subcutaneous administration of a positive comparator, Kineret(Anakinra)
Pharmacodynamics in comparison with Kineret(Anakinra): IL-6 inhibition assay | 1 day
  To explore pharmacodynamics in comparison with subcutaneous administration of a positive comparator, Kineret(Anakinra)

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong Ki Lee, Professor, Principal Investigator — Clinical Trial Center, Seoul National University Hospital
Locations (1):
- HANDOK Inc., Seoul, South Korea